CLINICAL TRIAL: NCT06424574
Title: The Effect of Motivational Interviewing on Hypoglycemia Fear Caring Failure and Self-commission in Parents of Children With Type 1 Diabetes
Brief Title: The Effect of Motivational Interviewing in Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Dilek Çiftci Baykal, assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DBAYKAL1421
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Motivational Interviewing; Type 1 Diabetes; Hypoglycemia; Fatigue; Self-Compassion
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Fatigue | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental): I. Interview: -Research for parents information was given about. Pretest forms were applied.
  Pre-test forms from filling;
  1. st interview after 2 weeks (45 min)
  2. nd interview after 2 weeks (45 min)
  3. Interviews after 2 weeks (45 min)
  4. th interview after 2 weeks (45 min)
  5. th interview: Post-test data were obtained 2 weeks after the last interview they were.
  Interventions: Behavioral: motivational interview
- Standard care (No Intervention): I. Interview: -Research for parents information was given about. Pretest forms were applied.
  II interview: Post-test data were obtained 2 weeks after the last interview they were.
  Post-test data were obtained 10 weeks after the last interview (it was ensured that the same time period passed with the experimental group)

INTERVENTIONS:
Behavioral: motivational interview — The sample of the second phase of the study consisted of 74 parents with Type 1 diabetes children, 37 of which were in the study group and 37 in the control group. İn the collection of data process, "Descriptive Information Form", "University of Virginia Parent Low Blood Sugar Scale", "BAKAS Care-Giving Impact Scale", "Fatigue Severity Scale", "Parental Version Of The Diabetes-Specific Self-Compassion Scale SCS-(Dp)" was used. The scales were applied at the beginning of the study and 10 weeks after the first data. After the first test data were obtained from each parent in our research group, four face-to-face motivational interviews were conducted at two-week intervals. In the xvii interviews, attempts were made to change and improve the behaviors and skills that parents felt inadequate within the scope of fear of hypoglycemia, caregiving, fatigue and self-compassion.
  Other Names: Experimental
  Arms: Motivational interviewing

SUMMARY:
This research was conducted in a randomized controlled experimental way to determine the effect of motivational interviewing on hypoglycemia fear, caregiving, fatigue and self-compassion in parents of children with Type 1 diabetes. The research was conducted with the parents of the patients who came to the Pediatric Endocrinology polyclinic of the Van Training and Research Hospital of the University of Health Sciences between July 26, 2021 and August 19, 2022. The research was carried out in two stages. The first stage was carried out methodologically to determine the validity and reliability of the "Parental Version Of The Diabetes-Specific Self-Compassion Scale SCS-(Dp)" in Turkish. The sample of the study was composed of 102 parents and the data were collected with the "Descriptive Information Form" and the " Parental Version Of The Diabetes-Specific Self-Compassion Scale SCS-(Dp)". "Language", "scope" and "construct" validity analyzes were used to evaluate the validity of the scale. KMO and Bartlett's Tests and factor analysis were evaluated for construct validity. As a result of the reliability analysis the Cronbach Alpha coefficient of the scale was found to be 0.817. As a result it was seen that the two 19 item sub-dimensions of the Turkish form of the "Parental Version Of The Diabetes Specific Self-Compassion Scale SCS-(Dp)" were confirmed for the Turkish form in the same way. The sample of the second phase of the study consisted of 74 parents with Type 1 diabetes children, 37 of which were in the study group and 37 in the control group. İn the collection of data process, "Descriptive Information Form", "University of Virginia Parent Low Blood Sugar Scale", "BAKAS Care-Giving Impact Scale", "Fatigue Severity Scale", "Parental Version Of The Diabetes-Specific Self-Compassion Scale SCS-(Dp)" was used.

DETAILED DESCRIPTION:
This research was conducted in a randomized controlled experimental way to determine the effect of motivational interviewing on hypoglycemia fear, caregiving, fatigue and self-compassion in parents of children with Type 1 diabetes. The research was conducted with the parents of the patients who came to the Pediatric Endocrinology polyclinic of the Van Training and Research Hospital of the University of Health Sciences between July 26, 2021 and August 19, 2022. The research was carried out in two stages. The first stage was carried out methodologically to determine the validity and reliability of the "Parental Version Of The Diabetes-Specific Self-Compassion Scale SCS-(Dp)" in Turkish. The sample of the study was composed of 102 parents and the data were collected with the "Descriptive Information Form" and the " Parental Version Of The Diabetes-Specific Self-Compassion Scale SCS-(Dp)". "Language", "scope" and "construct" validity analyzes were used to evaluate the validity of the scale. KMO and Bartlett's Tests and factor analysis were evaluated for construct validity. As a result of the reliability analysis the Cronbach Alpha coefficient of the scale was found to be 0.817. As a result it was seen that the two 19 item sub-dimensions of the Turkish form of the "Parental Version Of The Diabetes Specific Self-Compassion Scale SCS-(Dp)" were confirmed for the Turkish form in the same way. The sample of the second phase of the study consisted of 74 parents with Type 1 diabetes children, 37 of which were in the study group and 37 in the control group. İn the collection of data process, "Descriptive Information Form", "University of Virginia Parent Low Blood Sugar Scale", "BAKAS Care-Giving Impact Scale", "Fatigue Severity Scale", "Parental Version Of The Diabetes-Specific Self-Compassion Scale SCS-(Dp)" was used.

The scales were applied at the beginning of the study and 10 weeks after the first data. After the first test data were obtained from each parent in our research group, four face-to-face motivational interviews were conducted at two-week intervals. In the interviews, attempts were made to change and improve the behaviors and skills that parents felt inadequate within the scope of fear of hypoglycemia, caregiving, fatigue and self-compassion.

ELIGIBILITY:
Inclusion Criteria

* with a child diagnosed with T1D between the ages of 2-18 years,
* Can read and write Turkish, can be reached and communicated with,
* Orientation and co-operation,
* Without hearing, understanding and vision problems,
* Parents who agreed to participate in the study

Exclusion Criteria

* Communication difficulties,
* It is determined as being illiterate.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
The effect of motivational interviewing on parents' fear of hyperglycaemia Diabetes-Specific Self-Compassion Scale SCS-(Dp) | 13 monts
  University of Virginia Parental Fear of Low Blood Sugar Scale (P-LBSS)" It was developed by Gonder-Frederick and colleagues to assess parents' fear of their children's HG . The scale is a 4-point Likert-type scale consisting of 25 questions and two subscales (behavior, anxiety). Scoring on the scale is between 0 and 100, and the higher the score obtained from the scale, the higher the rate of HG fear increase. The Cronbach alpha reliability coefficients of the original scale were found to be 0.89, 0.76, and 0.91 for the total scale, behavior subscale, and anxiety subscale, respectively.
The effect of motivational interviewing on parents' caregiving effects | 13 months
  "Bakas Caregiving Impact Scale" is a measurement tool developed by Bakas and colleagues in 1999 to evaluate how the experiences of caregivers change with the caregiving process.The scale consists of a total of 15 items and shows positive and negative effects. The scale is a Likert-type scale, scored from +3 (in the best direction) to -3 (in the worst direction), ranging from 1 to 7. Scoring is done as -3=1, -2=2, -1=3, 0=4, +1=5, +2=6, +3=7. The lowest score that can be obtained from the scale is 15; the highest score is 10. As the scores increase, they are interpreted as ''change in the good direction'', and as the scores decrease, they are interpreted as ''change in the bad direction''. The internal consistency number of the original scale was found as 0.90, and the test-retest reliability was found as 0.81.
The effect of motivational interviewing on parents' fatigue severity | 13 months
  The Fatigue Severity Scale, which was also developed in the USA, was used for the first time in patients with multiple sclerosis. was used. Turkish validity and reliability study of the scale. It was conducted by Armutlu et al. in 2007. The scale has 9 questions and each question consists of 7 points. An increase in the scale score indicates an increase in the level of fatigue. The scale determines the fatigue status of individuals in the last 1 month. The questions are scored as strongly disagree (1)- strongly agree (7). The scale score is the average value of the questions. If the average score is 4 and above, it is considered as "severe fatigue". The lower the total score, the less "fatigue".
The effect of motivational interviewing on parents' level of self-compassion | 13 months
  The scale was developed by Tanenbaum et al. in 2020 to measure whether they have self-efficacy in coping with diabetes and coping with their emotions. The scale consists of 19 items and is a 5-point Likert-type scale (1="Almost never" and 5="Almost always"). Scale Positive dimension It has a two-factor structure as negative and negative dimension. The total score is calculated by averaging all items. Higher scores indicate higher diabetes-specific self-compassion

CONTACTS AND LOCATIONS:
Overall Officials: Dilek ÇİFTCİ BAYKA, Study Director — Yuzuncu Yil University
Locations (1):
- Van YUZUNCU YIL UNIVERSITY, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnard K, Thomas S, Royle P, Noyes K, Waugh N. Fear of hypoglycaemia in parents of young children with type 1 diabetes: a systematic review. BMC Pediatr. 2010 Jul 15;10:50. doi: 10.1186/1471-2431-10-50. PMID 20633252
- [Background] Channon S, Smith VJ, Gregory JW. A pilot study of motivational interviewing in adolescents with diabetes. Arch Dis Child. 2003 Aug;88(8):680-3. doi: 10.1136/adc.88.8.680. PMID 12876161
- [Background] Channon SJ, Huws-Thomas MV, Rollnick S, Hood K, Cannings-John RL, Rogers C, Gregory JW. A multicenter randomized controlled trial of motivational interviewing in teenagers with diabetes. Diabetes Care. 2007 Jun;30(6):1390-5. doi: 10.2337/dc06-2260. Epub 2007 Mar 10. PMID 17351283